CLINICAL TRIAL: NCT07150533
Title: Synergistic Effects of Green Tea Extract and Ginger Supplementation on Endurance Performance and Thermal Perception in Normal and Cold Environments: A Randomized Crossover Trial
Brief Title: Green Tea Extract and Ginger
Acronym: Thermal effect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Responsible Party: Principal Investigator, Süleyman Ulupınar, Associate Professor of Exercise Physiology, Erzurum Technical University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: ETU-Green Tea and Ginger
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Nutritional Supplementation; Exercise Physiology
MeSH Terms: interventions — Tea; ginger extract

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo Arm (Placebo Comparator): Participants receive a placebo consisting of maltodextrin in capsule form, matched in appearance and taste to the active supplements.
  Interventions: Dietary Supplement: Placebo Arm
- Green Tea Extract Arm (Experimental): Participants receive 500 mg of standardized green tea extract in capsule form.
  Interventions: Dietary Supplement: Green Tea Extract
- Ginger Arm (Experimental): Participants receive 1 g of ginger supplement in capsule form.
  Interventions: Dietary Supplement: Ginger
- Combined Supplement Arm (Experimental): Participants receive a combination of 500 mg green tea extract and 1 g ginger, both administered in capsule form.
  Interventions: Dietary Supplement: Combined Supplement (Green Tea + Ginger)

INTERVENTIONS:
Dietary Supplement: Placebo Arm — Participants receive a placebo consisting of maltodextrin in capsule form, matched in appearance and taste to the active supplements.
  Arms: Placebo Arm
Dietary Supplement: Green Tea Extract — Participants receive 500 mg of standardized green tea extract in capsule form.
  Arms: Green Tea Extract Arm
Dietary Supplement: Ginger — Participants receive 1 g of ginger supplement in capsule form.
  Arms: Ginger Arm
Dietary Supplement: Combined Supplement (Green Tea + Ginger) — Participants receive a combination of 500 mg green tea extract and 1 g ginger, both administered in capsule form.
  Arms: Combined Supplement Arm

SUMMARY:
This study investigates the effects of green tea extract and ginger supplementation, both individually and in combination, on endurance performance, metabolism, thermal comfort, and muscle soreness in recreationally active young men. Participants will complete cycling tests under both normal room temperature (21-24°C) and cold (5-7°C) conditions. The study uses a randomized, double-blind, placebo-controlled, crossover design to compare the outcomes of placebo, green tea, ginger, and combined supplementation. The findings may help to identify nutritional strategies that improve exercise performance and comfort in different environmental conditions.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, crossover trial is designed to evaluate the effects of green tea extract and ginger supplementation, both individually and in combination, on endurance performance, metabolic responses, thermal sensation, and muscle soreness in recreationally active men.

Sixteen healthy participants will complete eight experimental conditions: placebo, green tea extract (500 mg), ginger (1 g), and a combination of both, tested under normal (21-24°C) and cold (5-7°C) environments. Each condition will be separated by a washout period to avoid carryover effects.

Endurance capacity will be measured using a time-to-exhaustion cycling test at 70% of maximal oxygen uptake (VO₂max). Metabolic responses will be assessed by gas analysis to determine respiratory exchange ratio (RER). Perceptual measures will include the Borg Rating of Perceived Exertion (RPE) and a thermal sensation scale, while muscle soreness will be evaluated 24 hours post-exercise using a visual analog scale (VAS).

The study aims to determine whether the combined intake of green tea and ginger provides synergistic benefits over individual supplementation, particularly in cold environments where thermoregulation and endurance capacity are challenged. Findings may contribute to practical nutritional strategies that enhance exercise performance, comfort, and recovery under environmental stress conditions.

ELIGIBILITY:
Inclusion Criteria:

Male participants aged 18-35 years

Recreationally active (≥3 aerobic exercise sessions per week, ≥30 minutes per session, for at least 6 months)

VO₂max between 40-50 mL/kg/min (recreationally active fitness level)

Body mass index within the normal to slightly overweight range (approximately 18.5-27.5 kg/m²)

Willingness to comply with study requirements, including supplementation and exercise testing protocols

Provided written informed consent

Exclusion Criteria:

History of cardiovascular, respiratory, metabolic, or neurological disorders

Allergy or intolerance to green tea, ginger, or maltodextrin

Current use of ergogenic supplements, medications affecting metabolism, or stimulants (e.g., beta-blockers, caffeine pills)

Smoking or excessive alcohol consumption (>14 units per week)

Inconsistent exercise habits (<3 sessions/week in the past 6 months)

Participation in another clinical trial within the past 3 months

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Time to Exhaustion (TTE) | Immediately during each exercise test session (after supplement ingestion, under normal and cold environmental conditions)
  Endurance performance assessed as the total time in seconds participants are able to maintain cycling at 70% of VO₂max on a cycle ergometer, until volitional exhaustion defined as the inability to sustain a cadence of 60 rpm for 10 consecutive seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Technical University Sport Sciences Faculty, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Demirli A, Ulupinar S, Terzi M, Ozbay S, Ozkara AB, Gencoglu C, Ouergui I, Ardigo LP. Synergistic Effects of Green Tea Extract and Ginger Supplementation on Endurance Performance and Thermal Perception in Normothermic and Cold Environments: A Randomized, Placebo-Controlled, Double-Blind Crossover Trial. Nutrients. 2025 Sep 13;17(18):2949. doi: 10.3390/nu17182949. PMID 41010475